CLINICAL TRIAL: NCT03866382
Title: A Phase II Study of Ipilimumab, Cabozantinib, and Nivolumab in Rare Genitourinary Cancers (ICONIC)
Brief Title: Testing the Effectiveness of Two Immunotherapy Drugs (Nivolumab and Ipilimumab) With One Anti-cancer Targeted Drug (Cabozantinib) for Rare Genitourinary Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-01266; NCI-2019-01266 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A031702 (Other: Alliance for Clinical Trials in Oncology); A031702 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Bladder Adenocarcinoma; Bladder Clear Cell Adenocarcinoma; Bladder Mixed Adenocarcinoma; Bladder Neuroendocrine Carcinoma; Bladder Small Cell Neuroendocrine Carcinoma; Bladder Squamous Cell Carcinoma; Chromophobe Renal Cell Carcinoma; Collecting Duct Carcinoma; Invasive Bladder Giant Cell Urothelial Carcinoma; Invasive Bladder Lymphoepithelioma-Like Carcinoma; Invasive Bladder Nested Urothelial Carcinoma; Invasive Bladder Plasmacytoid Urothelial Carcinoma; Invasive Bladder Sarcomatoid Urothelial Carcinoma; Invasive Bladder Urothelial Carcinoma; Kidney Medullary Carcinoma; Large Cell Neuroendocrine Carcinoma; Malignant Testicular Leydig Cell Tumor; Malignant Testicular Sertoli Cell Tumor; Metastatic Bladder Carcinoma; Metastatic Bladder Clear Cell (Glycogen-Rich) Urothelial Carcinoma; Metastatic Bladder Giant Cell Urothelial Carcinoma; Metastatic Bladder Large Cell Neuroendocrine Carcinoma; Metastatic Bladder Lipid-Rich Urothelial Carcinoma; Metastatic Bladder Micropapillary Urothelial Carcinoma; Metastatic Bladder Plasmacytoid Urothelial Carcinoma; Metastatic Bladder Sarcomatoid Urothelial Carcinoma; Metastatic Bladder Small Cell Neuroendocrine Carcinoma; Metastatic Bladder Squamous Cell Carcinoma; Metastatic Chromophobe Renal Cell Carcinoma; Metastatic Kidney Medullary Carcinoma; Metastatic Malignant Genitourinary System Neoplasm; Metastatic Papillary Renal Cell Carcinoma; Metastatic Penile Carcinoma; Metastatic Prostate Small Cell Neuroendocrine Carcinoma; Metastatic Sarcomatoid Renal Cell Carcinoma; Metastatic Urethral Carcinoma; Papillary Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma; Stage IV Bladder Cancer AJCC v8; Stage IV Penile Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IV Urethral Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8; Urachal Adenocarcinoma; Urethral Clear Cell Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Urogenital Neoplasms; Penile Neoplasms; Urethral Neoplasms; Prostatic Neoplasms; Urachal adenocarcinoma | interventions — Specimen Handling; cabozantinib; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabozantinib, nivolumab, ipilimumab) (Experimental): Patients receive cabozantinib PO QD on days 1-21 of cycles 1-4 and on days 1-28 of subsequent cycles. Patients also receive nivolumab IV over 30 minutes on day 1 and ipilimumab IV over 90 minutes on day 1 of cycles 1-4. Patients then receive nivolumab IV over 30 minutes on day 1 of subsequent cycles. Treatment repeats every 21 days for cycles 1-4 and every 28 days for subsequent cycles for 2 years in the absence of disease progression or unacceptable toxicity. Patients may undergo echocardiography during screening and undergo CT or MRI, bone scan and blood and urine sample collection throughout the trial and may undergo PET/CT throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Procedure: Computed Tomography — Undergo CT and/or PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II trial studies how well cabozantinib works in combination with nivolumab and ipilimumab in treating patients with rare genitourinary (GU) tumors that has spread from where it first started (primary site) to other places in the body. Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cabozantinib, nivolumab, and ipilimumab may work better in treating patients with genitourinary tumors that have no treatment options compared to giving cabozantinib, nivolumab, or ipilimumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of cabozantinib s-malate (cabozantinib) combined with nivolumab and ipilimumab in the first or second-line (and beyond) setting for patients within each of the rare genitourinary (GU) variant histology group of interest, as measured by objective response rate (ORR).

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) for patients treated with cabozantinib combined with nivolumab and ipilimumab within each rare variant histology.

II. To estimate the overall survival (OS) for patients treated with cabozantinib combined with nivolumab and ipilimumab within each rare variant histology.

III. To estimate the clinical benefit rate (defined as complete response [CR] or partial response [PR] or stable disease [SD]) for patients treated with cabozantinib combined with nivolumab and ipilimumab within each rare variant histology.

IV. To assess the safety of treating patients with rare variant histologies with cabozantinib combined with nivolumab and ipilimumab.

V. To support tissue banking and collection of clinical follow-up data for GU tract rare histological variants.

EXPLORATORY OBJECTIVE:

I. To assess effects of treatment in patients with bone-only disease by bone scan.

OUTLINE:

Patients receive cabozantinib orally (PO) once daily (QD) on days 1-21 of cycles 1-4 and on days 1-28 of subsequent cycles. Patients also receive nivolumab intravenously (IV) over 30 minutes on day 1 and ipilimumab IV over 90 minutes on day 1 of cycles 1-4. Patients then receive nivolumab IV over 30 minutes on day 1 of subsequent cycles. Treatment repeats every 21 days for cycles 1-4 and every 28 days for subsequent cycles for 2 years in the absence of disease progression or unacceptable toxicity. Patients may undergo echocardiography during screening and undergo computed tomography (CT) or magnetic resonance imaging (MRI), bone scan and blood and urine sample collection throughout the trial and may undergo positron emission tomography (PET)/CT throughout the trial.

After completion of study treatment, patients are followed up every 2 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic disease defined as new or progressive lesions on cross-sectional imaging or bone scan. Patients must have at least:

  * One measurable site of disease as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1
  * One bone lesion on bone scan (tec99 or sodium fluoride [NaF] PET/CT, CT or MRI) for the bone-only cohort.
  * Histologically confirmed diagnosis of one of the following metastatic cohorts:

    * Small cell/ neuroendocrine carcinoma of the bladder (Cohort A)- All urothelial carcinomas with any amount of neuroendocrine differentiation (including small cell differentiation) will be included. If the tumor is purely neuroendocrine, metastasis from another site of origin should be clinically excluded
    * Adenocarcinoma of the bladder, or urachal adenocarcinoma, or bladder/urethra clear cell adenocarcinoma (Cohort B) - must be pure (per World Health Organization [WHO] definition), (i.e. urothelial carcinoma with glandular differentiation is not considered a pure adenocarcinoma
    * Squamous cell carcinoma of the bladder (Cohort C) - must be pure (i.e. urothelial carcinoma with squamous differentiation is not considered a pure squamous cell carcinoma)
    * Plasmacytoid urothelial carcinoma (Cohort D) - Tumor should show predominantly > or equal ~ 50% plasmacytoid histology (including all types of discohesive growth, such as tumors with signet-ring and/or rhabdoid features as well)
    * Any penile cancer (Cohort E)
    * Sarcomatoid renal cell carcinoma (Cohort F) - Tumor should be predominantly sarcomatoid ~ 50% (including rhabdoid differentiation) is also unclassified renal cell carcinomas (RCCs): all (assuming they are high grade with metastasis) malignant angiomyolipomas are allowed
    * Other miscellaneous histologic variants of the urothelial carcinoma, such as, but not limited to (Cohort G) : Micropapillary (Tumor should show predominantly > or equal 50% micropapillary architecture), giant cell, lipid-rich, clear cell and nested variants (Tumor should predominantly > or equal 50% show these features), large cell neuroendocrine carcinoma, lymphoepithelioma-like carcinoma and mixed patterns will be considered, as well as small cell neuroendocrine prostate cancer (Only treatment-naïve primary small cell of prostate with any amount of small cell component allowed. Post-treatment small cell prostatic carcinomas are not allowed), Malignant testicular Sertoli or Leydig cell tumors, and papillary and chromophobe RCC

      * Note: Translocation positive renal cell carcinoma patients are eligible. However, AREN1721 should be considered before this trial
    * Sarcomatoid urothelial carcinoma (Cohort H) - Tumor should show predominantly ~ 50% sarcomatoid differentiation
    * Renal medullary carcinoma (Cohort I) - Per World Health Organization (WHO) definition, ideally confirmed with immunostains
    * Bone-only metastatic GU tumors (non-prostate) (Cohort J) - All genitourinary histologies, except prostate are eligible
    * Renal Collecting Duct Carcinoma (Cohort K) - Per WHO definition (medullary involvement, predominant tubular morphology, desmoplastic stromal reaction, high grade cytology, infiltrative growth pattern, and absence of other renal cell carcinoma subtype or urothelial carcinoma)
    * Urethra carcinoma (Cohort L) - May be of any histology but if urothelial carcinoma then must be isolated to the urethra and not have metachronous or synchronous urothelial carcinoma of the bladder
  * H&E slides from diagnostic tumor tissue for retrospective central pathology review
* Patients may have received up to 2 systemic anti-cancer treatments or be treatment naive. Patients with small cell carcinoma should have received a platinum-based combination regimen either as neoadjuvant, adjuvant or first-line treatment). Patients in the bone-only cohort may be urothelial carcinoma histology but must receive standard cisplatin-based chemotherapy (if cisplatin-eligible)
* Age >= 18 years
* Patients must be able to swallow oral formulation of the tablets
* Karnofsky performance status >= 80%
* Absolute neutrophil count (ANC) >= 1,000/mcL
* Platelet count >= 75,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN). For subjects with known Gilbert's disease or similar syndrome with slow conjugation of bilirubin, total bilirubin =< 3.0 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3.0 x institutional upper limit of normal (ULN) (or =< 5 x ULN for patients with liver metastases or Gilbert's disease)
* Creatinine =< 1.5 x upper limit of normal (ULN) OR creatinine clearance >= 40 mL/min/1.73 m^2 (calculated using the Chronic Kidney Disease Epidemiology [CKD-EPI] equation or Cockcroft-Gault formula) for patients with creatinine levels above institutional normal
* Hemoglobin >= 9 g/dL (transfusion of packed red blood cells [PRBCs] allowed)
* Serum albumin >= 3.2 g/dL
* Lipase and amylase =< 2.0 x ULN and no radiologic (on baseline anatomical imaging) or clinical evidence of pancreatitis
* Prior treatment with MET or VEGFR inhibitors is allowed. However, prior cabozantinib will not be allowed. Also, patients that have received both prior MET or VEGF and prior PD-1/PD-L1/CTLA-4 (sequentially or in combination) are also not allowed
* No prior treatment with any therapy on the PD-1/PD-L1 axis or anti- CTLA-4/CTLA-4 inhibitors with the exception of patients with "urothelial carcinoma" histology (cohorts D, H, J, L)
* Human immunodeficiency virus (HIV)-positive patients are eligible if on stable dose of highly active antiretroviral therapy (HAART), no clinically significant drug-drug interactions are anticipated with the current HAART regimen, CD4 counts are greater than 350 and viral load is undetectable
* Patients with rheumatoid arthritis and other rheumatologic arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication only and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies etc. are eligible but should be considered for rheumatologic evaluation for the presence of target organ involvement and potential need for systemic treatment
* Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones or medications (e.g. thyroiditis managed with propylthiouracil [PTU] or methimazole) including physiologic oral corticosteroids are eligible
* Patients who have evidence of active or acute diverticulitis, intra-abdominal abscess, and gastrointestinal (GI) obstruction, within 12 months are not eligible
* Women of childbearing potential must have a negative pregnancy test =< 7 days prior to registration

  * Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Post menopause is defined as amenorrhea >= 12 consecutive months. Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason
* Pregnant women may not participate in this study because with cabozantinib, nivolumab, and ipilimumab have potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cabozantinib, nivolumab, and ipilimumab, breastfeeding should be discontinued if the mother is treated with these agents
* The patient has received no cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 2 weeks before the first dose of study treatment
* The patient has received no radiation therapy:

  * To the lungs and mediastinum or abdomen within 4 weeks before the first dose of study treatment, or has ongoing complications, or is healing from prior radiation therapy
  * To brain metastasis within 3 weeks for whole-brain radiotherapy (WBXRT), and 2 weeks for stereotactic body radiation therapy (SBRT) before the first dose of study treatment
  * To the abdomen within 4 weeks before the first dose of study treatment, or has ongoing complications, or is healing from prior radiation therapy
  * To any other site(s) within 2 weeks before the first dose of study treatment
* The patient has received no radionuclide treatment within 6 weeks of the first dose of study treatment
* The patient has received no prior treatment with a small molecule kinase inhibitor within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment
* The patient has received no prior treatment with hormonal therapy within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment. Subjects receiving gonadotropin-releasing hormone (GnRH) agonists and antagonists are allowed to participate
* The patient has not received any other type of investigational agent within 14 days before the first dose of study treatment
* The patient must have recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from toxicity due to all prior therapies except alopecia, neuropathy and other non-clinically significant adverse events (AEs) defined as lab elevation with no associated symptoms or sequelae
* The patient may not have active brain metastases or epidural disease. Patients with brain metastases previously treated with whole brain radiation or radiosurgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible. Neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 3 months before starting study treatment. Baseline brain imaging with contrast-enhanced CT or MRI scans for subjects with known brain metastases is required to confirm eligibility
* No concomitant treatment with warfarin. Aspirin (up to 325 mg/day), thrombin or factor Xa inhibitors, low-dose warfarin (=< 1 mg/day), prophylactic and therapeutic low molecular weight heparin (LMWH) are permitted
* No chronic concomitant treatment with strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort) or strong CYP3A4 inhibitors

  * Because the lists of these agents are constantly changing, it is important to regularly consult medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* The patient has not experienced any of the following:

  * Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood per day within 1 months before the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The patient has no tumor invading any major blood vessels
* The patient has no evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib. Patients with rectal tumor masses are not eligible
* The patient has no uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening.
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
    * The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before randomization. Note: if initial QTcF is found to be > 500 ms, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is =< 500 ms, the subject meets eligibility in this regard
    * Any history of congenital long QT syndrome
    * Any of the following within 6 months before registration of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias (patients with atrial fibrillation are eligible)
      * Stroke (including transient ischemic attack [TIA], or other ischemic event)
      * Myocardial infarction
      * Cardiomyopathy
  * No significant gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following that have not resolved within 28 days before the first dose of study treatment:

      * Active peptic ulcer disease
      * Acute diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or malabsorption syndrome
    * None of the following within 2 years before the first dose of study treatment:

      * Abdominal fistula or genitourinary fistula
      * Gastrointestinal perforation
      * Bowel obstruction or gastric outlet obstruction
      * Intra-abdominal abscess. Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 2 years before the first dose of study treatment
  * Disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement are not eligible
  * No other clinically significant disorders such as:

    * Severe active infection requiring IV systemic treatment within 14 days before the first dose of study treatment
    * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
    * History of organ or allogeneic stem cell transplant
    * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment (for asymptomatic patients with an elevated thyroid-stimulating hormone [TSH], thyroid replacement may be initiated if clinically indicated without delaying the start of study treatment)
  * No history of major surgery as follows:

    * Major surgery within 3 months of the first dose of cabozantinib; however, if there were no wound healing complications, patients with rapidly growing aggressive cancers, may start as soon as 6 weeks if wound has completely healed post-surgery
    * Minor surgery within 1 month of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications excluding core biopsies and mediport placement
    * Complete wound healing from prior surgery must be confirmed before the first dose of cabozantinib irrespective of the time from surgery
* No history of severe hypersensitivity reaction to any monoclonal antibody
* No evidence of active malignancy, requiring systemic treatment within 2 years of registration
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib, nivolumab, ipilimumab or other agents used in study
* No positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection. If HBV sAG is positive, subsequent ribonucleic acid (RNA) polymerase chain reaction (PCR) must be negative
* No patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. These include, but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 5 years
  An objective response is defined as a confirmed complete response (CR) or partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. A confirmed tumor response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. Will be estimated by the number of confirmed objective responses divided by the total number of evaluable patients. Confidence intervals for the true ORR will be calculated.

SECONDARY OUTCOMES:
Duration of response | From time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 years
  Defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented.
Progression-free survival (PFS) | From start of treatment to time of progression or death, whichever occurs first, assessed up to 5 years
  The median its 95% confidence interval will be determined and will be summarized using the Kaplan-Meier estimator.
Overall survival | Up to 5 years
  The median its 95% confidence interval will be determined and will be summarized using the Kaplan-Meier estimator.
Clinical benefit rate (CBR) | Up to 5 years
  A confirmed clinical benefit is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart or a confirmed stable disease at two consecutive tumor assessments at least 3 months apart. The CBR will be estimated by the number of patients with confirmed clinical benefit divided by the total number of evaluable patients. Confidence intervals for the true CBR will be calculated using exact binomial confidence intervals.
Incidence of adverse events (AE) | Up to 5 years
  Will be assessed using Common Terminology Criteria for Adverse Events version 5.0. The maximum of a particular AE will be determined for each patient. Tables will summarize the number and relative frequency of patients observing an AE as well as the number and relative frequency of patients experiencing any AE of grade 3 or greater.

OTHER OUTCOMES:
Effects of treatment in patients with bone-only disease | Up to 5 years
  The bone-only tumor patients will be evaluated in an exploratory fashion (if no RECIST measurements are available). A maximum of 15 patients with bone-only disease will be enrolled and evaluated using PFS for a descriptive analysis of the effect of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (576):
- United States (575):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Rush MD Anderson Cancer Center at Rush Oak Park, Oak Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Freeman Physician Group of Pittsburg, Pittsburg, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University Cancer Specialists - Alcoa, Alcoa, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Pan American Center for Oncology Trials LLC, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Girardi DM, Niglio SA, Mortazavi A, Nadal R, Lara P, Pal SK, Saraiya B, Cordes L, Ley L, Ortiz OS, Cadena J, Diaz C, Bagheri H, Redd B, Steinberg SM, Costello R, Chan KS, Lee MJ, Lee S, Yu Y, Gurram S, Chalfin HJ, Valera V, Figg WD, Merino M, Toubaji A, Streicher H, Wright JJ, Sharon E, Parnes HL, Ning YM, Bottaro DP, Cao L, Trepel JB, Apolo AB. Cabozantinib plus Nivolumab Phase I Expansion Study in Patients with Metastatic Urothelial Carcinoma Refractory to Immune Checkpoint Inhibitor Therapy. Clin Cancer Res. 2022 Apr 1;28(7):1353-1362. doi: 10.1158/1078-0432.CCR-21-3726. PMID 35031545